CLINICAL TRIAL: NCT05452850
Title: Longitudinal Changes in Left and Right Ventricular Global Strain After Chemotherapy in Cardiac Light Chain Amyloidosis: Prognostic Significance
Brief Title: Longitudinal Changes in Left and Right Ventricular Global Strain After Chemotherapy in Cardiac Light Chain Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Mutlu, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 2021-53809
Record Dates: First submitted 2022-07-02; First posted 2022-07-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Amyloid Cardiomyopathy; Congestive Heart Failure; Chemotherapy Effect
Keywords: Cardiac amyloidosis; Cardiomyopathy; Heart failure; Chemotherapy; Echocardiography; Strain imaging
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Light Chain Cardiac Amyloidosis: Participants with light chain cardiac amyloidosis actively receiving chemotherapy or undergoing autologous bone marrow transplant
  Interventions: Diagnostic Test: Left and Right Ventricular Global Strain Imaging

INTERVENTIONS:
Diagnostic Test: Left and Right Ventricular Global Strain Imaging — Two-dimensional, color Doppler, spectral Doppler, and 3D digital echocardiographic image recordings will be taken from parasternal, apical, subcostal, and modified sections using a Philips Epiq CVx echocardiography device and X5-1 probe. Conventional parameters, additional parameters, and strain analyzes will be performed with speckle tracking echocardiography from these recordings.
  Other Names: TomTec AutoStrain Suite Software; Philips Epiq CVx Echocardiography System; Philips X5-1 3D Echocardiography Probe

SUMMARY:
The purpose of this study to assess the longitudinal changes in left and right ventricular global strain after chemotherapeutic strategies in cardiac light chain amyloidosis.

DETAILED DESCRIPTION:
Light chain amyloidosis is a disease characterized by localized or systemic accumulation of amyloid fibrils in tissues caused by abnormal folding of light chain immunoglobulins and affecting organ functions. In the treatment, chemotherapeutic agents are used that prevent the clonal proliferation of plasma cells in the bone marrow. Although the hematological response is standardized in evaluating the treatment response, there is no adequately effective method for assessing cardiac response. Despite the use of various scores, imaging-based systems continue to be developed to increase the sensitivity of these methods.

After being informed about the study, it is planned to recruit and follow-up AL-Amyloidosis patients with cardiac involvement who are currently receiving/planned chemotherapy followed by hematology or who are planned for bone marrow transplantation within 1 year after obtaining written consent from the patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients who give the informed consent
* Patients with cardiac primary light chain amyloidosis or due to multiple myeloma who are newly diagnosed, currently receiving chemotherapeutic treatment, or are scheduled for bone marrow transplantation

Exclusion Criteria:

* A history of myocardial infarction, coronary artery disease, PCI and revascularization
* < 18 years old
* A history of severe aortic and mitral valve disease
* Patients who do not give the informed consent
* A history of severe hypertension (SBP>180 mmHg or DBP ≥110 mmHg or the need to use three or more antihypertensive agents)
* Stable coronary artery patients with ischemia data in stress tests (exertion test, myocardial perfusion scintigraphy)
* Presence of non-amyloidosis, systemic, inflammatory or autoimmune disease
* Patients whose cardiac imaging is not interpretable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-90 years with cardiac primary light chain amyloidosis or due to multiple myeloma who are newly diagnosed, currently receiving chemotherapeutic treatment, or are scheduled for bone marrow transplantation will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The longitudinal changes in left and right ventricular global strain after chemotherapy in cardiac light chain amyloidosis | Change from Baseline left and right ventricular global strain at 1 year
  In this study, the effects of treatment strategies on left and right ventricular global and regional strain and its relationship with mortality and morbidity will be investigated in patients with AL-amyloidosis, who are still under treatment, and newly diagnosed with AL-amyloidosis.

SECONDARY OUTCOMES:
Evaluation of the effects of treatment strategies on other cardiac morphological and functional changes in standard echocardiographic imaging | Baseline, and 1st, 3rd, 6th, 12th Month follow-up
  Evaluation of the effects of treatment strategies on other cardiac morphological and functional changes in standard echocardiographic imaging was planned as a secondary objective.

CONTACTS AND LOCATIONS:
Overall Officials: Burçak Kılıçkıran Avcı, Assoc Prof., Study Chair — Istanbul University - Cerrahpasa; Deniz Mutlu, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sperry BW, Ikram A, Hachamovitch R, Valent J, Vranian MN, Phelan D, Hanna M. Efficacy of Chemotherapy for Light-Chain Amyloidosis in Patients Presenting With Symptomatic Heart Failure. J Am Coll Cardiol. 2016 Jun 28;67(25):2941-8. doi: 10.1016/j.jacc.2016.03.593. PMID 27339491
- [Result] Witteles RM, Liedtke M. AL Amyloidosis for the Cardiologist and Oncologist: Epidemiology, Diagnosis, and Management. JACC CardioOncol. 2019 Sep 24;1(1):117-130. doi: 10.1016/j.jaccao.2019.08.002. eCollection 2019 Sep. PMID 34396169
- [Result] Bak M, Kim D, Choi JO, Kim K, Kim SJ, Jeon ES. Prognostic Implication of Longitudinal Changes of Left Ventricular Global Strain After Chemotherapy in Cardiac Light Chain Amyloidosis. Front Cardiovasc Med. 2022 Jun 24;9:904878. doi: 10.3389/fcvm.2022.904878. eCollection 2022. PMID 35811735